CLINICAL TRIAL: NCT06654219
Title: Protective Benefits of a Clear Liquid Diet on Residual Gastric Content in Patients Taking Glucagon Like Peptide-1 Receptor Agonist Prior to Anesthesia
Brief Title: Protective Benefits of a Clear Liquid Diet on Residual Gastric Content in Patients Taking Glucagon Like Peptide-1 Receptor (GLP-1 RA) Agonist Prior to Anesthesia
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Sudipta Sen, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: HSC-MS-24-0940
Record Dates: First submitted 2024-10-21; First posted 2024-10-23 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Pulmonary Aspiration
Keywords: Glucagon Like Peptide-1 Receptor (GLP-1 RA); full stomach

STUDY DESIGN:
Who Masked: Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- GLP-1 RA users with prolonged fasting instructions (Experimental)
  Interventions: Other: GLP-1 RA users with prolonged fasting instructions
- GLP-1 RA users with standard NPO instructions (Active Comparator)
  Interventions: Other: GLP-1 RA users with standard NPO instructions

INTERVENTIONS:
Other: GLP-1 RA users with prolonged fasting instructions — NPO for solids: 24 hours prior to procedure, clear liquid diet (CLD) for 24 hours with last intake of clears no less than 2 hours prior to a procedure.GLP-1 RA will not be held prior to surgery and usual dosing schedule will be followed prior to procedure.
  Arms: GLP-1 RA users with prolonged fasting instructions
Other: GLP-1 RA users with standard NPO instructions — NPO after midnight prior to procedure; Minimum solid fasting duration of 8 hours for solids and 2 hours for liquids. Last dose of GLP-1 RA no less than 7 days prior to procedure.
  Arms: GLP-1 RA users with standard NPO instructions

SUMMARY:
The purpose of this study is to determine if prolonged fasting from solids and transitioning to a CLD for 24 hours is protective to decrease RGC in patients on GLP-1 RAs presenting for upper endoscopy, to determine if prolonged fasting is associated with increased thirst, hunger and anxiety, To determine if signs and symptoms of nausea, vomiting, retching, abdominal bloating, and abdominal pain are present on the day of surgery, to see if there is any variability between preoperative gastric ultrasound assessment and volume of gastric contents visualized on upper endoscopy, to determine time of gastric emptying by serial Gastric ultrasonography (GUS) scans every 2 hours in subjects who presented with an initial at-risk scan, to determine the choice of anesthesia used based on preoperative GUS results, to determine if there were any adverse events recorded in this study group, to determine if duration of GLP-1 RA therapy has an association with residual gastric content (RGC). and to determine if dosing of GLP-1 RA has an association with RGC.

ELIGIBILITY:
Inclusion Criteria:

* Patients taking Glucagon Like Peptide-1 Receptor (GLP-1 RA) agonists
* Undergoing upper endoscopy only - no colonoscopy due to prep

Exclusion Criteria:

* Previous gastric resection or bypass
* Gastric band in situ
* Previous fundoplication
* Large hiatal hernia
* Pregnant patients
* Recent trauma
* Inability to turn to the right lateral decubitus position.
* Patients on erythromycin, metoclopramide, domperidone, opioids.
* Gastroparesis previous

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 136 (Estimated)
Dates: Start 2025-10-30 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Number of participants that show prevalence of increased RGC determined using preoperative GUS | prior to procedure ( within 2 hours before procedure)
  Participants with increased RGC will have solids, thick fluid, or clear fluids >1.5ml/kg in the gastric antrum in the right lateral decubitus position

SECONDARY OUTCOMES:
Number of participants that show thirst as assessed by the VAS | prior to procedure ( within 2 hours before procedure)
  This is measured in a linear scale from 1-10, higher number showing worse outcome
Number of participants that show hunger as assessed by the VAS | prior to procedure ( within 2 hours before procedure)
  This is measured in a linear scale from 1-10, higher number showing worse outcome
Number of participants that show anxiety as assessed by the VAS | prior to procedure ( within 2 hours before procedure)
  This is measured in a linear scale from 1-10, higher number showing worse outcome

CONTACTS AND LOCATIONS:
Overall Officials: Sudipta Sen, MD, FASA, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No